CLINICAL TRIAL: NCT03193398
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy And Safety Study Of BTRX-246040 Administered Once Daily In Patients With Major Depressive Disorder With Or Without Anhedonia
Brief Title: BTRX-246040 Administered Once Daily to Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEP-MDD-201
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Anhedonia; antidepressant; Nociceptin; NOPR
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTRX-246040 (Experimental): 40 mg administered orally as 1 capsule QD for 1 week, followed by 80 mg as 2 capsules QD for 7 weeks.
  Interventions: Drug: BTRX-246040 oral capsule(s)
- Placebo (Placebo Comparator): administered orally as 1 capsule QD for 1 week, followed by 2 capsules QD for 7 weeks.
  Interventions: Drug: Placebo oral capsule(s)

INTERVENTIONS:
Drug: BTRX-246040 oral capsule(s) — BTRX-246040 administered once daily to patients with MDD for 8 weeks
  Arms: BTRX-246040
Drug: Placebo oral capsule(s) — administered once daily to patients with MDD for 8 weeks
  Arms: Placebo

SUMMARY:
This study will determine the efficacy, safety, and tolerability of a once-daily (QD) dose of up to 80 mg of BTRX-246040 for 8 weeks in participants with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of MDD as defined by DSM-5 criteria and have had at least 1 prior major depressive episode in the past 10 years
* Patients must present with a new current episode of MDD and the duration of the current episode must be at least 4 weeks but not longer than 18 months.
* At Visit 1 (screening) and Visit 2 (baseline), patients must have clinically significant depressive symptoms defined by tandem (investigator- and computer-administered) Montgomery-Asberg Depression Rating Scale (MADRS) total scores ≥ 26 with a difference of ≤ 7 points between the Investigator- and computer-administered MADRS total scores
* Patients must have a CGI-S score ≥ 4 at Visit 2 (baseline).

Exclusion Criteria:

* Patients who present with any current DSM-5 disorder other than MDD which is the focus of treatment.
* Patients who are homicidal in the opinion of the Investigator or are at suicidal risk (any suicide attempts within 12 months prior to Visit 1 [screening] or any suicidal intent, including a plan, within 3 months prior to Visit 1 [screening]; C-SSRS answer of "YES" on item 4 or 5 [suicidal ideation]; Investigator- or computer-administered MADRS score of ≥ 5 on item 10 [suicidal thoughts]; by Investigator clinical evaluation).
* Patients cannot have any history of substance or alcohol use disorder within 12 months prior to Visit 1 (screening) per DSM-5 criteria
* Patients must not have a clinically significant comorbid disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Tiller, MD, Study Director — BlackThorn Therapeutics, Inc.
Locations (8):
- United States (8):
  - United States, Cerritos, California
  - United States, Garden Grove, California
  - United States, Florida, Jacksonville, Florida
  - United States, Lauderhill, Florida
  - United States, Florida, Orlando, Florida
  - United States, Libertyville, Illinois
  - United States, Rochester, New York
  - United States, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 104 subjects were randomized for the study NEP-MDD-201
Period: Overall Study
Arm/Group | BTRX-246040 | Placebo
Started | 53 | 51
Completed | 38 | 35
Not Completed | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTRX-246040 | Placebo | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.29) | 42.6 (15.00) | 40.9 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 43 | 41 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  Black or African American | 22 | 19 | 41
  Native Hawaiian or Other Pacific Islanders | 0 | 1 | 1
  White | 24 | 26 | 50
  Multiracial | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Investigator-administered MADRS Total Score From Baseline BTRX-246040 and Placebo
Description: The Investigator-administered MADRS includes 10 items assessing the following symptoms: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (absence of symptom) to 6 (severe symptom); the overall score ranges from 0 to 60. MADRS total scores from 0 to 6 indicate normal/symptom absent, from 7 to 19 indicate mild depression, from 20 to 34 indicate moderate depression, and from 35 to 60 indicate severe depression.
Time Frame: Week 8
Population: The full analysis set (FAS) contained all patients in the randomized set who received at least 1 dose of study medication and had at least 1 post-dose efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | -15.0 (1.73) | -13.6 (1.79)
Statistical Analysis 1: Comparison: BTRX-246040 vs Placebo; Difference in LS Means (BTRX-246040 - Placebo); Test type: Other; p = 0.5939, MMRM; MMRM: mixed model for repeated measures; Mean Difference (Net) = -1.3, 95% CI 2-sided [-6.3 to 3.6]

2. Secondary Outcome: Change From Baseline in Investigator-administered MADRS-6 Total Score
Description: The Investigator-administered MADRS-6 subscale focuses on the core symptoms of depression and assesses the following symptoms: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts. Each item is scored from 0 (absence of symptom) to 6 (severe symptom); the overall score ranges from 0 to 36. The change from baseline in the Investigator-administered MADRS-6 subscale was analyzed using the same method as the MADRS efficacy endpoint, substituting the baseline MADRS-6 subscale as the covariate in place of the MADRS total score.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | -10.7 (1.17) | -9.7 (1.21)
Statistical Analysis 1: Comparison: Placebo; Analysis of Change from Baseline in Investigator-administered MADRS-6 Total Score at week 8; Test type: Other; p = 0.5503, MMRM; MMRM: mixed model for repeated measures; Mean Difference (Net) = -1.0, 95% CI 2-sided [-4.4 to 2.3]

3. Secondary Outcome: Change From Baseline in Investigator-administered HADS-A (Hospital Anxiety and Depression Scale - Anxiety Subscale) Score
Description: The Investigator-administered Hospital Anxiety and Depression Scale (HADS) subscales comprises of 7 questions regarding Depression and 7 questions regarding Anxiety. Each question is rated on a scale from 0 - 3. The outcome of the HADS questionnaire is two total scores, the HADS-A (for anxiety) and the HADS-D (for depression). Both total scores are graded on a scale of 0 - 21 and can be categorized as Normal (0 - 7), Borderline Abnormal (8 - 10) and Abnormal (11 - 21). Higher scores indicate higher levels of anxiety and depression.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | -2.6 (0.67) | -3.5 (0.70)
Statistical Analysis 1: Comparison: BTRX-246040 vs Placebo; Test type: Other; p = 0.3906, MMRM; MMRM: mixed model for repeated measures; Mean Difference (Net) = 0.8, 95% CI 2-sided [-1.1 to 2.8]

4. Secondary Outcome: Change From Baseline in Investigator-administered HADS-D (Hospital Anxiety and Depression Scale - Depression Subscale) Score
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | -5.0 (0.76) | -5.9 (0.80)
Statistical Analysis 1: Comparison: BTRX-246040 vs Placebo; Test type: Other; p = 0.4187, MMRM — +/-; MMRM: mixed model for repeated measures; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.3 to 3.1]

5. Secondary Outcome: Change From Baseline in Investigator-administered Dimensional Anhedonia Rating Scale (DARS)
Description: The Investigator-administered Dimensional Anhedonia Rating Scale (DARS) is a 17-item questionnaire with each answer between 0 and 4 on a Likert scale grading (0=Not at all, 1=Slightly, 2=Moderately, 3=Mostly, 4=Very Much). Therefore, the DARS total score is on a scale of 0 - 68. The DARS Total score is broken down into four dimensions; Hobbies, Food/Drink, Social Activities and Sensory Experience.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | 13.7 (16.7) | 2.91 (3.04)
Statistical Analysis 1: Comparison: BTRX-246040 vs Placebo; Test type: Other; p = 0.4869, MMRM; MMRM: mixed model for repeated measures; Mean Difference (Net) = -3.0, 95% CI 2-sided [-11.5 to 5.5]

6. Secondary Outcome: Change From Baseline in Investigator-administered Snaith-Hamilton Pleasure Scale (SHAPS) Score
Description: The Investigator-administered Snaith Hamilton Pleasure Scale (SHAPS) is a 14-item questionnaire. The SHAPS is scored two different ways. Under the original scoring method, each question has 4 responses, 2 of which imply agreement (Definitely Agree, Agree; each scored as 0) and 2 which imply disagreement (Disagree, Strongly Disagree; each scored as 1). Therefore, the SHAPS total score ranges 0 - 14. In this study, in addition to the traditional scoring method, an alternative scoring method will assign 1 - Strongly Agree, 2 - Agree, 3 - Disagree, and 4 - Strongly Disagree. Using this alternative scoring method, the total score ranges 14-56. In both scoring systems, higher scores indicate greater anhedonia.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | BTRX-246040 | Placebo
Number analyzed (Participants) | 52 | 50
Change in score on a scale from baseline | -6.7 (1.24) | -7.9 (1.28)
Statistical Analysis 1: Comparison: BTRX-246040; Test type: Other; p = 0.5178, MMRM; MMRM: mixed model for repeated measures; Mean Difference (Net) = 1.2, 95% CI 2-sided [-2.4 to 4.7]

ADVERSE EVENTS:
Time Frame: Up to week 10
Arm/Group | BTRX-246040 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/51
Other Adverse Events (participants affected / at risk) | 34/53 | 27/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTRX-246040 (N=53) | Placebo (N=51)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTRX-246040 (N=53) | Placebo (N=51)
Headache (Nervous system disorders) | 8 | 13
Somnolence (Nervous system disorders) | 3 | 7
Dizziness (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Disturbance In Attention (Nervous system disorders) | 0 | 1
Formication (Nervous system disorders) | 0 | 1
Hypogeusia (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 3 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 0 | 2
Dermatitis Infected (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Irritability (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 2 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 2
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2
Amylase Increased (Investigations) | 0 | 1
Lipase Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1
Vision Blurred (Eye disorders) | 2 | 0
Eyelid Oedema (Eye disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Benign Ethnic Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hot Flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03193398/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03193398/SAP_001.pdf